CLINICAL TRIAL: NCT00798174
Title: The Effect of an Azygos Vein Coil on Defibrillation Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0045
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: DFT; Congestive Heart failure (CHF); ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single group undergoing crossover in therapy (defibrillation testing with two different device configurations).
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard configuration vs. azygos coil (Experimental): The DFT with the standard Superior Vena Cava (SVC) coil vs. DFT with the azygos coil.
  In this crossover study, each patient serves and own control, with defibrillation testing performed with and with the azygos coil
  Interventions: Device: Standard configuration vs. azygos coil

INTERVENTIONS:
Device: Standard configuration vs. azygos coil — Addition of an azygos vein defibrillation coil instead of a standard SVC coil.
  Other Names: Medtronic 6937A Lead

SUMMARY:
When implantable cardiac defibrillators are implanted (ICDs), the defibrillation threshold (DFT), of the amount of energy required to effectively terminate life-threatening arrhythmias is determined. The device is then programmed to discharge a larger amount of energy in order to provide a safety margin. In some patients, the DFT is so high, that an adequate safety margin is not programmable. Placement of a defibrillation lead in the azygos vein has been found to be helpful in these patients. This goal of this trial is to attempt to quantify the average reduction in the DFT (if any) that results from the addition of the azygos lead.

DETAILED DESCRIPTION:
Patients undergoing placement of an ICD for the primary or secondary prevention of sudden cardiac death will be asked to participate. Patients will undergo implantation of a standard right ventricular ICD lead at the time of ICD implantation. In addition, patient will receive another high voltage ICD lead placed in the azygos vein as has been previously described in the literature (1). After sedating the patient, the DFT will be determined using a binary search algorithm. This consists of testing the device at a given output for the first shock after inducing ventricular fibrillation (VF). Should the shock fail, external defibrillation will be attempted, as is the standard method for performing DFT testing. As per the standard method of DFT testing, VF will be induced a second time, with the shock strength dependent on the success of the first shock. If the first shock was unsuccessful, the second will be at a higher output. If the first shock was successful, the second will be at a lower output. A third shock will then be delivered, based on the success or failure of the preceding shock to define the DFT. Of note, as the device can be programmed to give multiple shocks for one episode, VF will not necessarily need to be induced each time. For example, VF could be induced, and the device programmed to give a 20 Joule (J) shock followed by a 23J shock if not successful, thus limiting the number of VF inductions required. DFT testing will be done using both the standard configuration of high voltage leads as well as using the azygos lead. We hypothesize that using the azygos lead will result in a lower DFT.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing elective placement of an ICD for the primary or secondary prevention of sudden cardiac death is eligible. Exclusion criteria include any contraindication to endovascular ICD implantation which includes but is not limited to; active infection, occluded venous access, or inability to perform DFT testing secondary to the inability to sedate the patient or hemodynamic compromise.

Exclusion Criteria:

* Any contraindication to ICD or the inability to place an azygos vein coil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2009-11-18 (Actual); Study Completion 2009-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W. Smith, DPhil, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Cooper JA, Latacha MP, Soto GE, Garmany RG, Gleva MJ, Chen J, Faddis MN, Smith TW. The azygos defibrillator lead for elevated defibrillation thresholds: implant technique, lead stability, and patient series. Pacing Clin Electrophysiol. 2008 Nov;31(11):1405-10. doi: 10.1111/j.1540-8159.2008.01203.x. PMID 18950297
- [Background] Cesario D, Bhargava M, Valderrabano M, Fonarow GC, Wilkoff B, Shivkumar K. Azygos vein lead implantation: a novel adjunctive technique for implantable cardioverter defibrillator placement. J Cardiovasc Electrophysiol. 2004 Jul;15(7):780-3. doi: 10.1046/j.1540-8167.2004.03649.x. PMID 15250862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing Implantable Cardioverter-Defibrillator (ICD) implantation in the electrophysiology laboratory were recruited. Both outpatients (recruited from the electrophysiology clinic) and inpatients (recruited from Barnes-Jewish Hospital) were included.
Groups:
- Standard Configuration First: 1. st time period (approx. 0.5 hour): Defibrillation Threshold (DFT) testing was performed with standard configuration first. A maximum of three inductions of ventricular fibrillation (VF) with defibrillation were performed to establish a standard configuration threshold. There were at least 5 minutes between defibrillation tests, so the standard configuration period was approximately 0.5 hour.
  2. nd time period: The azygos coil was then added for the second phase.
  (Azygos vein coil: Addition of an azygos vein defibrillation coil in place of a standard superior vena cava (SVC) coil.)
- Azygos Coil Configuration First: 1. st time period (approx 0.5 hr): DFT testing was performed with an azygos coil in place first. A maximum of three inductions of VF with defibrillation were performed to establish a standard configuration threshold. There were at least 5 minutes between defibrillation tests, so the standard configuration period was approximately 0.5 hour.
  2. nd time period (approx 0.5 hour): The azygos coil was then excluded from the shocking configuration and replaced by the standard SVC coil configuration for the second phase.
Period: Overall Study
Arm/Group | Standard Configuration First | Azygos Coil Configuration First
Started | 16 | 16
Completed | 12 | 13
Not Completed | 4 | 3
Not completed — inability to implant azygos coil | 3 | 3
Not completed — Inability to sedate for DFT testing | 1 | 0

BASELINE CHARACTERISTICS:
Population: 32 patients were enrolled. There was inability to place an and azygos coil in 6. 1 could not be sedated for defibrillation testing. 25 patients were analyzed.
Groups:
- Standard SVC Coil vs. Azygos Coil: The DFT with the standard SVC coil vs. DFT with the azygos vein coil in place.
  Azygos vein coil: Addition of an azygos vein defibrillation coil instead of a standard SVC coil.
Arm/Group | Standard SVC Coil vs. Azygos Coil
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Difference in the DFT With an Azygos Vein Coil Versus the Standard SVC Coil.
Description: Defibrillation threshold will be estimated by repeat defibrillation testing using an azygos coil and using an SVC coil (and compared).
  The outcome measure quoted below is the mean DFT using the azygos coil vs. the mean DFT using the standard configuration.
Time Frame: During the course of the implant procedure and testing
Population: All enrolled patient who were able to undergo azygos coil implant and defibrillation testing.
Measure: Mean (Standard Deviation); unit: Joules
Groups:
- Standard Configuration vs. Azygos Coil: The DFT with the standard SVC coil vs. DFT with the azygos coil. In this crossover study, each patient serves and own control, with defibrillation testing performed with and with the azygos coil
  Standard configuration vs. azygos coil: Addition of an azygos vein defibrillation coil instead of a standard SVC coil.
Arm/Group | Standard Configuration vs. Azygos Coil
Number analyzed (Participants) | 25
Joules
  DFT wtih Azygos coil | 10.4 (7.7)
  DFT with Standard Configuration | 12.2 (8.61)
Statistical Analysis 1: Comparison: Standard Configuration vs. Azygos Coil; The null hypothesis is that there is no difference between the DFT using the azygos coil vs. the standard configuration. Paired t-test (two-tailed), used due to construction of study with DFT determined in both configurations in each patient, yields p=0.103; Test type: Superiority — The null hypothesis was that the azygos coil does not reduce the DFT. (A reduced DFT is superiority); p = 0.103, t-test, 2 sided — Threshold for significance is 0.05; Paired t-test

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Definitions are as the clinicaltrials.gov definitions.
  Patients were follow for clinically for 24 hours after their implant and defibrillation testing procedure.
Groups:
- Standard Configuration vs. Azygos Coil Configuation: The DFT with the standard SVC coil vs. DFT with the azygos vein coil in place.
  Since all subjects underwent attempted azygos vein implantation, the implantation procedure was the same for the arm in which the standard configuration was tested first and the arm in which the azygos configuration was tested. first. Therefore, the two arms (Standard configuration tested first and Azygos configuration tested first) were combined for the purpose of adverse events.
Arm/Group | Standard Configuration vs. Azygos Coil Configuation
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Configuration vs. Azygos Coil Configuation (N=25)
Loss of intergrity of Lead introducer (Blood and lymphatic system disorders) | 1 (1) — In one patient with very constricted vascular access, the introducer sheath for azygos vein lead became torn. Small fragments remained embedded in the soft tissue near the access site. No sequelae and no prolongation of hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes